CLINICAL TRIAL: NCT06404190
Title: DIODE LASER PHOTOACTIVATION OF 3% HYDROGEN PEROXIDE FOR POCKET DECONTAMINATION A CLINICAL STUDY
Brief Title: Diode Laser Photo Activation for Pocket Reduction Decontamination A Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KCDSHEC/IP/2023/P11
Record Dates: First submitted 2024-04-10; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pocket, Periodontal; Periodontal Inflammation; Periodontal Attachment Loss; Periodontitis
MeSH Terms: conditions — Periodontal Pocket; Periodontal Attachment Loss; Periodontitis | interventions — Lasers, Semiconductor; Hydrogen Peroxide

STUDY DESIGN:
Intervention Model Description: GROUP A: ultrasonic GROUP B: laser and hydrogen peroxide
Masking Description: GROUP A: 10 SRP ALONE GROUP B: 10 SRP+3%HYDROGEN PEROXIDE+DIODE LASER
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DIODE LASER PHOTOACTIVATION OF 3% HYDROGEN-PEROXIDE FOR POCKET DECONTAMINATION - A CLINICAL STUDY (Experimental): 1)To evaluate the effectiveness of 3% hydrogen peroxide as an adjunct to scaling and root planning with diode laser irriadation 2. To compare the clinical and microbiology outcome of SRP + 3% hydrogen peroxide + diode laser and SRP alone
  Interventions: Combination Product: Diode laser and 3% hydrogen peroxide

INTERVENTIONS:
Combination Product: Diode laser and 3% hydrogen peroxide — Hydrogen peroxide due to its super radicals has a local antimicrobial effect. Since hydrogen peroxide can be easily available in a clinical setting and is cost-effective. It could be used for photo disinfection along with lasers.
  The diode lasers that belong to the 655-980 nm spectrum could represent a safer alternative. Because of the transmission or scattering effect on hydroxyapatite, diode lasers have no effect on hard tissues and deposits. The photoactivation procedure uses photolysis of hydrogen peroxide with 810nm laser.
  Hydrogen peroxide acts as an endogenous dye, which can increase the laser effect at this level and also generate ROS. Thus the combination of 3% H2O2 and laser light generate hydroxyl radicals as a result of photoactivation.
  Therefore, the diode laser stimulation of 3%hydrogen peroxide has been utilized adjunctive to SRP to optimize clinical outcomes.

SUMMARY:
Routine non surgical periodontal thearpy often fails to achieve complete elimination of pathogenic microorganism. This could be attiributable to deep periodontal pockets, root concavities, furcation involvement etc. Systemic and local antimicrobials have been used adjunctively with scaling and root planning to optimize the results. They have their own draw backs namely antibiotic resistance and narrow spectrum of action over periodontal pathogens. In the last decade lasers applications have diversified occupying greater part of the periodontal treatment strategies. Photodynamic thearpy has shown conflicting results as a adjunctive thearpy. The routinely used dyes are Methyelene blue, indocyanine green and rose bengal .These dyes are difficult to procure and may not be economical . Hydrogen peroxide due to its super radicals has a local antimicrobial effect. Since hydrogen peroxide can be easily available in a clinical setting and is cost effective. It could be used for photodisinfection . From the near-infrared spectrum lasers, the Nd-YAG laser can remove periodontal pathogens because of its thermal effect. However, changes in the neighboring tissues can be attributed to these unwanted thermal effects. The diode lasers that belong to the 655-980 nm spectrum could represent a safer alternative.Because of the transmission or scattering effect on hydroxyapatite, diode lasers have no effect on calculus. Anaerobic bacterial species intermedia produce black pigments in Brucella media from blood agar. Hemoglobin in the soft periodontal tissues behaves like a chromophore, being absorbed by the diode laser. Photoactivated procedure use photolysis of hydrogen peroxide with 810nm laser. It acts as an endogenous dye, which can increase the laser effect at this level and also generate ROS stopped immediately after the laser irridation. Therefore, the diode laser stimulation of 3%hydrogen peroxide has been utilized adjuvantive to SRP to optimize clinical outcome.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled single-blind clinical trial to assest the antimicrobial effect of non surgical periodontal thearpy with SRP alone , and photoactivation of 3% H2O2 with 810nm diode in combination with SRP. Based on the method of randomization, each patient was allocated to one of the two treatment groups as follows: Group 1: SRP as monotherapy; Group 2: SRP+H2O2photoactivation with diode laser. One week after the baseline periodontal examination and microbiological sampling, scaling and root planning is carried out using conventional ultrasonic scaler .Every patient received oral hygiene instructions that included modified BASS brushing technique . In Group 1- Only SRP: Group 2- 3% H2O2solution was inserted to the bottom of the periodontal pocket using a disposable plastic needle similar to the endodontic irrigation followed by diode 810 nm laser irridation with 1.1 W, continuous wave (CW) with 300mm The activated fiber was applied from the bottom to the free gingival margin of the periodontal pocket in parallel with the root surface and side-to-side movements were performed for*30 sec per test surface. Microbiological assessment was performed 1 week before periodontal treatment.

Microbiological samples were obtained from the selected periodontal pockets at baseline (before treatment) and at 1 month after the periodontal treatment by the examiner. Sterile paper points will be placed into periodontal pocket to collect the gcf sample for 30 sec, then it is transfer to Eppendorf tubes(individual sampling) having (thioglycate broth) and incubated for 2 hrs then broth is( vortex). Later sample is cultured on the anerobic blood agar media and incubated in gas jar with anerobic gas pack for 48hrs and colony counting is done after 48hrs of incubation. Clinical periodontal parameters PPD, BOP, CAL and mobility were assessed baseine and 3 months after the periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years of age Minimum of 5mm of periodontal probing depth Patient under going orthodontic prosthodontic restorative treatment Stage 2 and 3 Grade B and C periodontitis acc to 2017 classification

Exclusive Criteria:

Pregnacy systemic disease people

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Probing pocket Depth | 3 months
  1. Probing pocket Depth (PPD), dept measuring from cej to depth of pocket through william probe

SECONDARY OUTCOMES:
DIODE LASER PHOTOACTIVATION OF 3% HYDROGEN-PEROXIDE FOR POCKET DECONTAMINATION - A CLINICAL STUDY | 3 month
  Colony count

CONTACTS AND LOCATIONS:
Locations (1):
- Anusha s, Bengaluru, Karnataka, India